CLINICAL TRIAL: NCT00704106
Title: HBV Viral Suppression by Entecavir in Adefovir Partial Responders
Brief Title: Hepatitis B Virus (HBV) Viral Suppression by Entecavir in Adefovir Partial Responders
Acronym: ADVPR
Status: Completed | Type: Observational
Sponsor: Pacific Health Foundation (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: PHF008
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Hepatitis B
Keywords: Hepatitis B; HBV; Treatment
MeSH Terms: conditions — Hepatitis B | interventions — entecavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1: Persistent viremia after 48 weeks or longer.
  Interventions: Drug: Entecavir
- Group 2: <2 log IU/mL drop from initial HBVDNA after 12 weeks of adefovir
  Interventions: Drug: Entecavir
- Group 3: Patients who responded to adefovir and were switched to entecavir.
  Interventions: Drug: Entecavir
- Group 4: Patients with 160 copies/mL (100 IU/mL) or higher at the time of medication switch.
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Entecavir — 0.5 or 1 mg dose qd
  Other Names: Baraclude

SUMMARY:
We propose a largely retrospective study with short-term prospective follow-up in a subgroup of patients who have not yet been treated with 48 weeks of entecavir following partial response to adefovir. The aim of the study is to describe sequential virologic response to adefovir and entecavir.

DETAILED DESCRIPTION:
Amendment was made, and approved by WIRB in January 2009, to this protocol: We propose a largely retrospective study with short-term prospective follow-up in a subgroup of patients who have not yet been treated with 96 weeks of entecavir following adefovir treatment. The aim of the study is to describe sequential virologic response to adefovir and entecavir.

ELIGIBILITY:
KEY INCLUSION CRITERIA:

* Age 18 years or older
* All genders and ethnicity
* Positive HBsAg
* HBeAg positive and negative
* Pretreatment HBV DNA of 10,000 copies/mL or higher (for purposes of this study, both copies and equivalent IU measurements will be recorded and analyzed)
* Patients who are switched to, or prescribed, entecavir after treatment with adefovir for at least 12 weeks by the providing physician.
* Patients with and without prior lamivudine exposure will be enrolled but enrollment of lamivudine experienced cases will be limited to no more than 30 patients total

KEY EXCLUSION CRITERIA:

* Patients who refused to consent to the study
* Patients younger than 18
* Vulnerable subjects such as pregnant women, prisoners, employees, patients with significant cognitive deficits.
* Patients with prior exposure to another nucleoside for more than 2 weeks. Those with prior exposure to lamivudine will be enrolled under conditions detailed above.
* HIV co-infection
* HCV co-infection
* HDV co-infection
* Recipients of solid organ transplantation
* Patients who receive high-dose steroid (60 mg/d or higher and for longer than 10 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Age 18 years or older
  * All genders and ethnicity
  * Positive HBsAg
  * HBeAg positive and negative
  * Pretreatment HBV DNA of 10,000 copies/mL or higher (for purposes of this study, both copies and equivalent IU measurements will be recorded and analyzed)
  * Patients who are switched to, or prescribed, entecavir after treatment with adefovir for at least 12 weeks by the providing physician
  * Patients with and without prior lamivudine exposure will be enrolled but enrollment of lamivudine experienced cases will be limited to no more than 30 patients total
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
HBV DNA PCR after 12 weeks of entecavir from the time of medication switching: percent of patients with <2log drop in HBV DNA and percent of patients with complete viral suppression during adefovir versus during entecavir. | 48 weeks or after

SECONDARY OUTCOMES:
HBV DNA PCR after 24 weeks of entecavir from the time of medication switching. | 48 weeks or after
HBV DNA PCR after 48 weeks of entecavir from the time of medication switching. | 48 weeks or after
BR and CR at 24 and 48 weeks of therapy with entecavir. | 48 weeks or after.
BR and CR for longer duration of therapy if available. | 48 weeks or after.

CONTACTS AND LOCATIONS:
Overall Officials: Huy N Trinh, M.D., Principal Investigator — Pacific Health Foundation; Mindie H Nguyen, M.D., M.A.S., Principal Investigator — Pacific Health Foundation
Locations (5):
- United States (5):
  - Stanford University Medical Center, Palo Alto, California
  - San Jose Gastroenterology, San Jose, California
  - Asian Village Medical Clinic, Chicago, Illinois
  - Houston Gastroenterology Clinic, Houston, Texas
  - Digestive Health Associates of Texas, Plano, Texas

REFERENCES:
- [Background] McMahon BJ. Epidemiology and natural history of hepatitis B. Semin Liver Dis. 2005;25 Suppl 1:3-8. doi: 10.1055/s-2005-915644. PMID 16103976
- [Background] Chen CJ, Yang HI, Su J, Jen CL, You SL, Lu SN, Huang GT, Iloeje UH; REVEAL-HBV Study Group. Risk of hepatocellular carcinoma across a biological gradient of serum hepatitis B virus DNA level. JAMA. 2006 Jan 4;295(1):65-73. doi: 10.1001/jama.295.1.65. PMID 16391218
- [Background] Iloeje UH, Yang HI, Su J, Jen CL, You SL, Chen CJ; Risk Evaluation of Viral Load Elevation and Associated Liver Disease/Cancer-In HBV (the REVEAL-HBV) Study Group. Predicting cirrhosis risk based on the level of circulating hepatitis B viral load. Gastroenterology. 2006 Mar;130(3):678-86. doi: 10.1053/j.gastro.2005.11.016. PMID 16530509
- [Background] Liaw YF, Sung JJ, Chow WC, Farrell G, Lee CZ, Yuen H, Tanwandee T, Tao QM, Shue K, Keene ON, Dixon JS, Gray DF, Sabbat J; Cirrhosis Asian Lamivudine Multicentre Study Group. Lamivudine for patients with chronic hepatitis B and advanced liver disease. N Engl J Med. 2004 Oct 7;351(15):1521-31. doi: 10.1056/NEJMoa033364. PMID 15470215
- [Background] Lok AS, McMahon BJ. Chronic hepatitis B. Hepatology. 2007 Feb;45(2):507-39. doi: 10.1002/hep.21513. No abstract available. PMID 17256718
- [Background] Keeffe EB, Dieterich DT, Han SH, Jacobson IM, Martin P, Schiff ER, Tobias H, Wright TL. A treatment algorithm for the management of chronic hepatitis B virus infection in the United States: an update. Clin Gastroenterol Hepatol. 2006 Aug;4(8):936-62. doi: 10.1016/j.cgh.2006.05.016. Epub 2006 Jul 14. PMID 16844425
- [Background] Shaw T, Locarnini S. Entecavir for the treatment of chronic hepatitis B. Expert Rev Anti Infect Ther. 2004 Dec;2(6):853-71. doi: 10.1586/14789072.2.6.853. PMID 15566330
- [Background] Chan HL, Heathcote EJ, Marcellin P, Lai CL, Cho M, Moon YM, Chao YC, Myers RP, Minuk GY, Jeffers L, Sievert W, Bzowej N, Harb G, Kaiser R, Qiao XJ, Brown NA; 018 Study Group. Treatment of hepatitis B e antigen positive chronic hepatitis with telbivudine or adefovir: a randomized trial. Ann Intern Med. 2007 Dec 4;147(11):745-54. doi: 10.7326/0003-4819-147-11-200712040-00183. Epub 2007 Oct 1. PMID 17909201
- [Background] Keeffe EB, Zeuzem S, Koff RS, Dieterich DT, Esteban-Mur R, Gane EJ, Jacobson IM, Lim SG, Naoumov N, Marcellin P, Piratvisuth T, Zoulim F. Report of an international workshop: Roadmap for management of patients receiving oral therapy for chronic hepatitis B. Clin Gastroenterol Hepatol. 2007 Aug;5(8):890-7. doi: 10.1016/j.cgh.2007.05.004. Epub 2007 Jul 13. PMID 17632041
- [Background] Colonno RJ, Rose R, Baldick CJ, Levine S, Pokornowski K, Yu CF, Walsh A, Fang J, Hsu M, Mazzucco C, Eggers B, Zhang S, Plym M, Klesczewski K, Tenney DJ. Entecavir resistance is rare in nucleoside naive patients with hepatitis B. Hepatology. 2006 Dec;44(6):1656-65. doi: 10.1002/hep.21422. PMID 17133475
- [Background] Tenney DJ, Rose RE, Baldick CJ, Pokornowski KA, Eggers BJ, Fang J, Wichroski MJ, Xu D, Yang J, Wilber RB, Colonno RJ. Long-term monitoring shows hepatitis B virus resistance to entecavir in nucleoside-naive patients is rare through 5 years of therapy. Hepatology. 2009 May;49(5):1503-14. doi: 10.1002/hep.22841. PMID 19280622
- [Background] Hadziyannis SJ, Tassopoulos NC, Heathcote EJ, Chang TT, Kitis G, Rizzetto M, Marcellin P, Lim SG, Goodman Z, Ma J, Arterburn S, Xiong S, Currie G, Brosgart CL; Adefovir Dipivoxil 438 Study Group. Long-term therapy with adefovir dipivoxil for HBeAg-negative chronic hepatitis B. N Engl J Med. 2005 Jun 30;352(26):2673-81. doi: 10.1056/NEJMoa042957. PMID 15987916
- [Background] Hadziyannis SJ, Tassopoulos NC, Heathcote EJ, Chang TT, Kitis G, Rizzetto M, Marcellin P, Lim SG, Goodman Z, Ma J, Brosgart CL, Borroto-Esoda K, Arterburn S, Chuck SL; Adefovir Dipivoxil 438 Study Group. Long-term therapy with adefovir dipivoxil for HBeAg-negative chronic hepatitis B for up to 5 years. Gastroenterology. 2006 Dec;131(6):1743-51. doi: 10.1053/j.gastro.2006.09.020. Epub 2006 Sep 20. PMID 17087951
- [Background] Ha NB, Ha NB, Garcia RT, Trinh HN, Vu AA, Nguyen HA, Nguyen KK, Levitt BS, Nguyen MH. Renal dysfunction in chronic hepatitis B patients treated with adefovir dipivoxil. Hepatology. 2009 Sep;50(3):727-34. doi: 10.1002/hep.23044. PMID 19517525
- [Derived] Nguyen NH, Trinh HN, Nguyen TT, Do ST, Tran P, Nguyen HA, Nguyen KK, Garcia RT, Lutchman GA, Nguyen MH. Safety and efficacy of entecavir in adefovir-experienced patients. J Gastroenterol Hepatol. 2015 Jan;30(1):43-50. doi: 10.1111/jgh.12728. PMID 25168842